CLINICAL TRIAL: NCT00485043
Title: Effects of Modified T'ai Chi Exercise on Physical Function, Pain, and Stiffness in Older Adults With Lower Extremity Osteoarthritis
Brief Title: Effects of Modified T'ai Chi on Symptoms in Older Adults With Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUMC-JCarpenter dissertation-1
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Osteoarthritis
Keywords: T'ai Chi; Osteoarthritis; Exercise; Older adults
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Modified T'ai Chi: T'ai Chi for Arthritis

SUMMARY:
The purpose of this study was to evaluate the effects of TC for Arthritis on physical function, pain, and stiffness in older adults with knee/hip OA. Two hypotheses were tested:

1. Individuals in the TC group will demonstrate greater improvements in physical function compared to control group participants.
2. Individuals in the TC group will demonstrate greater decreases in pain and stiffness compared to control group participants.

DETAILED DESCRIPTION:
Exercise is considered a vital component of osteoarthritis (OA) treatment. T'ai Chi (TC) is a unique exercise intervention with low-velocity movements. Few studies have addressed the effects of TC on arthritis symptoms and function. TC for Arthritis was modified specifically for people with OA and consists of a standardized set of forms.

The purpose of this study was to evaluate the effectiveness of a low-dose TC for Arthritis on physical function, pain, and stiffness in individuals with OA.

Twenty-seven older adults with OA (mean age-81.3 years) completed an 8 week non-randomized controlled pre-post test quasi-experimental design study of TC for Arthritis. Physical function, pain, and stiffness were measured at baseline and 8 weeks for the TC and control groups using the WOMAC™ 3.1 Index. Qualitative data from interviews and participant observations were analyzed in order to understand the participants' expectations and experiences with TC.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk independently,
* Speak and understand English,
* Understand the consent process; and
* Give informed consent.

Exclusion Criteria:

* Participation in rehabilitation or another TC class,
* At the time of recruitment; and
* Inability to confirm medical stability for safe participation with healthcare provider.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
physical function | 8 weeks

SECONDARY OUTCOMES:
pain and stiffness | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Teel S. Teel, BSN, PhD, Study Chair — University of Kansas Medical Center; Geraldine R. Neuberger, BSN, EdD, Study Chair — University of Kansas Medical Center